CLINICAL TRIAL: NCT06309849
Title: Efficacy of Physical Therapy Intervention in Cervical Angina Patients at Jerash University Office Employees, "Randomized Clinical Trail".
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ibrahim Abuzaid, Director, Head of Department of Physiotherapy for Cardiovascular/Respiratory and Geriatrics, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jerash University
Record Dates: First submitted 2024-02-10; First posted 2024-03-13 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Randomized Control Trail (RCT) will be used in the study. Participants will be dived into experimental group and control group. Each group will includes 30 participants.
Who Masked: Participant
Masking Description: includes 30 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efficacy of Physical Therapy Intervention in Cervical Angina Patients (Experimental): Randomized Control Trail (RCT) will be used in the study. Participants will be dived into experimental group and control group. Each group will includes 30 participants.The physiotherapy program intervention will includes cervical traction, cervical mobilization, Sub occipital release, Muscle energy technique. and ultra sound with parameters 5 min × 3 times × 4 weeks, 1 MHz, continuous: 1.5 W/cm2; pulsed: 2.5 W/cm2, for study group.
  Interventions: Other: Manual physiotherapy intervention( cervical traction, suboccipital release, muscle energy technique)
- know the effect of Physical Therapy Intervention in Cervical Angina Patients (Placebo Comparator): 30 participants in control.The physiotherapy program intervention will include ultrasound with parameters 5 min × 3 times × 4 weeks, 1 MHz, continuous: 1.5 W/cm2; pulsed: 2.5 W/cm2
  Interventions: Other: Manual physiotherapy intervention( cervical traction, suboccipital release, muscle energy technique)

INTERVENTIONS:
Other: Manual physiotherapy intervention( cervical traction, suboccipital release, muscle energy technique) — Manual physiotherapy intervention( cervical traction, suboccipital release, muscle energy technique) strengthening exercises for neck muscles, ultrasound with parameters 5 min × 3 times × 4 weeks, 1 MHz, continuous: 1.5 W/cm2; pulsed: 2.5 W/cm2.
  Other Names: Strengthening exercises for neck muscles, ultrasound with parameters 5 min × 3 times × 4 weeks, 1 MHz, continuous: 1.5 W/cm2; pulsed: 2.5 W/cm2,

SUMMARY:
Cervicogenic angina (CA) is defined as paroxysmal angina- like pain that originates from the disorders of the cervical spine or other neck structures. Because CA mimics typical cardiac angina, symptoms in the elderly with cervical spondylosis are more frequently misdiagnosed Nakajima H, 2006. Patients with CA may have suffered symptoms for longer periods of time and seen several clinicians due to conflicting cardiac exams. Clinicians and patients are unaware that CA symptoms are stemming from cervical spine disorders. However, the mechanism of pain occurrence in patients with CA remains unclear.

DETAILED DESCRIPTION:
Randomized Control Trail (RCT) will be used in the study. Participants will be divided into two groups (experimental and control groups). Each group will include 30 participants.

The study population will be employees working in JU from different departments.

A total of 60 participants will be included in the study. Their weight ranged from (50 kilograms) to (100 kilograms). And their height ranged from (150 centimeters) to (190 centimeters). And their body mass index ranged from (22.2) to (27.7). This will be divided into 2 groups with 30 participants in each group.

The data collected will focus on measuring the Range of Motion (ROM) of the cervical spine using an Electro-Goniometer, the pain using Visual Analogue Scale (VAS), and the Hart Rate (HR) using an electro cardio Graphic (ECG).

The study setting will be JU, located in Jerash City, Jordan.

ELIGIBILITY:
Inclusion Criteria:

* cervical spondylosis, cervical disc, cervical instability

Exclusion Criteria:

* Cardiovascular diseases ( ischemic heart disease, heart failure, valvular disease)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
1-Hart Rate (HR) (bpm) using Electro Cardiac Graphic (ECG). 2- Blood pressure (mm Hg) using Sphygmomanometer. | Four weeks
  1- Hart Rate (HR) (bpm) using Electro Cardiac Graphic (ECG). 2- Blood pressure (mm Hg) using 1-Hart Rate (HR) using Electro Cardiac Graphic (ECG). 2- Blood pressure using Sphygmomanometer.

SECONDARY OUTCOMES:
3- Range of Motion (ROM) (in degrees) of the cervical spine using Electro-Goniometer. 4- the pain using Visual Analogue Scale (VAS) from (0-10) | 4 Weeks
  3- Range of Motion (ROM) (in degrees) of the cervical spine using Electro-Goniometer. 4- the pain using Visual Analogue Scale (VAS) from ( 0-10)

IPD SHARING:
Plan to Share IPD: Yes
After publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication
Access Criteria: Not yet

REFERENCES:
- [Result] Chien JT, Hsieh MH, Yang CC, Chen IH, Lee RP. Anterior Cervical Discectomy and Fusion Versus Conservative Treatment for Cervical Angina Conservative Treatment. Clin Spine Surg. 2021 Nov 1;34(9):E514-E521. doi: 10.1097/BSD.0000000000001178. PMID 33828047